CLINICAL TRIAL: NCT04083794
Title: Exploration of Blood Flow Regulation to Bone in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, J. Andrew Taylor, Associate Chair for Research, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018P000156; R21AR074054-01A1 (NIH)
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Bone Blood Flow Regulation
Keywords: bone perfusion; bone blood flow regulation; vascular sympathetic activity; skeletal loading; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Head-Down Tilt

STUDY DESIGN:
Intervention Model Description: This is a Basic Experimental study with Humans with able-bodied individuals and individuals with spinal cord injury (SCI). This study is a cross sectional assessment and will have 1 or 2 visits consisting of 2 protocols where individuals will undergo several physical maneuvers during which bone perfusion response will be assessed. Protocol #1 will investigate tibial perfusion response to tibial loading. Protocol #2 will investigate tibial perfusion response to isometric handgrip exercise and tilt. Volunteers can choose to do one or both protocols during 1 or 2 laboratory visits.
  Study completion update: In able bodied adults, we have investigated tibial perfusion in response to isometric handgrip exercise, cold pressor test, leg dependency, reactive hyperemia, and sublingual nitroglycerin. In adults with spinal cord injury, we have investigated tibial perfusion in response to isometric handgrip exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laboratory based assessments (Other): The current study has no arms; it is a cross-sectional assessment where all participants will undergo the same procedures.
  Interventions: Other: Laboratory based assessments

INTERVENTIONS:
Other: Laboratory based assessments — physical maneuvers to assess physiological responses in bone blood flow
  Other Names: handgrip; tilt; tibial loading

SUMMARY:
Without blood flow, bone cannot maintain its integrity. Bone blood flow responds to various local and systemic factors, however, bone perfusion in humans remains relatively unstudied. The investigators will study key mechanisms that regulate bone perfusion in able-bodied and contrast responses to those with spinal cord injury (SCI). SCI is a model of chronic reduced loading with loss of sympathetic regulation. In tibial cortical bone, the investigators will: 1) determine the impact of compressive loading with and without muscle contractions; 2) determine the impact of vascular sympathetic activity and systemic perfusion pressure; 3) compare the response between able-bodied and those with SCI. Acute metabolic needs of bone due to loading increase flow substantially. In addition, the bone vasculature is innervated by a rich network of sympathetic nerves that serve a functional purpose in the control of blood flow. A critical limitation to the study of bone blood flow in humans has been the lack of non-invasive assessments. Previously, the investigators developed a near infrared spectroscopy (NIRS) device to non-invasively assess blood content in bone and assessed tibial perfusion in response to exercise. Here, the investigators will test the hypothesis that bone blood flow increases proportional to loading conditions in both able-bodied individuals and those with SCI. The investigators will also test the hypothesis that there are decreases in blood bone flow that are proportional to increases in leg vascular sympathetic outflow in the able-bodied, but that changes in bone blood flow are proportional to changes in blood pressure in those with SCI. The proposed research will be some of the first to determine the control of bone flow in humans.

DETAILED DESCRIPTION:
All tissues of the human body require adequate perfusion to provide oxygen and nutrients to meet metabolic demands. It has long been known that the arterial system in bone is of overwhelming importance and that without blood flow, bone cannot maintain its integrity. Indeed, there is an extensive network of arteries, arterioles, and capillaries that supply human bone. Moreover, blood flow to bone is responsive to various local and systemic factors that can determine the overall health of bone. However, bone perfusion in humans remains relatively unstudied and so the underlying mechanisms that regulate bone blood flow are not well understood. The investigators propose to study key mechanisms that regulate bone perfusion in able-bodied individuals and to contrast them with spinal cord injured (SCI) individuals. SCI represents a human 'model' of chronic reduced loading with loss of sympathetic regulation below the level of injury that likely alters control of bone perfusion. Accordingly, our aims are to: 1) Determine the impact of compressive loading with and without associated muscle contractions on tibial perfusion; 2) Determine the impact of vascular sympathetic activity and systemic perfusion pressure on tibial perfusion; 3) Compare the changes in tibial perfusion in response to local and systemic factors between able-bodied and those with SCI.

The majority of work in bone blood flow has been in animals and/or has focused on the association between adequate or inadequate perfusion and bone health. For example, inadequate flow has been associated with bone loss, impaired growth, and delayed fracture healing. However, the acute metabolic needs of bone due to loading either with or without associated muscle contractions increase flow substantially. Indeed, within two minutes of isolated muscle contractions alone, tibial perfusion has been shown to increase significantly. Furthermore, when there is compressive loading with associated muscle contractions, flow to bone can double. Similarly, skeletal unloading for as short as ten minutes cuts femoral perfusion by half. Although it is unclear what specific local factors (e.g., metabolic by-products) with loading might be responsible for regulation of blood flow, these data strongly suggest that perfusion to bone is highly responsive to skeletal loading. Indeed, it appears that similar regulatory mechanisms may be at play in control of flow to bone and skeletal muscle during exercise. In addition, the bone vasculature is richly innervated by sympathetic nerves. Application of norepinephrine decreases blood flow to both intact bone and isolated bone. Likewise, sympathetic stimulation decreases flow to bone via alpha-adrenergic receptor activation. Moreover, smooth muscle of arterioles in bone respond as expected to vasodilators and vasoconstrictors. Hence, sympathetic innervation of the bone vasculature serves a functional purpose in control of flow. If this were not the case, independent of the link between bone metabolism and bone flow, the arterial network in bone would act as a simple pressure passive system.

A critical limitation to the study of bone flow in humans has been the lack of noninvasive assessments. Thus, it has been difficult to elucidate the mechanisms that control perfusion to bone. The dense nature of bone makes it difficult to investigate perfusion and the techniques used to quantify circulation in other tissues are either difficult or impossible to apply to bone in vivo. the investigators recently demonstrated the efficacy of a near infrared spectroscopy (NIRS) system to non-invasively detect changes in hemoglobin content in the tibia. Although our preliminary work showed the utility of NIRS, it was not designed to provide insight to blood flow regulation and disentangle the various possible contributors to bone perfusion. Here the investigators propose to study different mechanisms that control blood flow to bone in both able-bodied and spinal cord injured (SCI). The SCI population will offer valuable insights to the mechanisms of perfusion as several contributors (i.e. loading and vascular sympathetic control) are either reduced or disrupted.

Study completion update: Given the exploratory nature of this study, the scope has been adjusted to address the challenges and limitations that have occurred during the duration of this research. Nonetheless the work completed has provided unprecedented findings on key mechanisms of vascular regulation in bone in vivo in humans. We were not able to assess the impact of compressive loading with or without associated muscle contractions on tibial perfusion due to marked impact of motion artefacts on the near infrared spectroscopy technology used to assess tibial perfusion. In young healthy adults, we have assessed the impact of vascular sympathetic activity (in response to two stimuli: isometric handgrip exercise and cold pressor test) and increased perfusion pressure (in response to two stimuli: leg dependency and reactive hyperemia). In those with spinal cord injury, given the inherent limitations of working with this population (i.e., increased spasticity, autonomic dysreflexia), we have assessed the impact of lack of vascular sympathetic activity on tibial blood flow regulation. Furthermore, we have extended the initial work and in young healthy adults we have investigated an additional key regulation mechanism of the tibial vasculature, namely nitric oxide mediated vasodilation.

Even though we have obtained data during compressive loading in both able-bodied and adults with spinal cord injury, the data were not usable due to motion artefacts. In addition, the data obtained in those with SCI during leg dependency and reactive hyperemia were insufficient or unusable (due to increased spasticity and autonomic dysreflexia) to draw any meaningful conclusions.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females
* individuals with spinal cord injuries, between 3 and 24 months post injury, with complete injuries according to the American Spinal Injury Association Impairment Scale A and B, with injuries at T6 and below

Exclusion Criteria:

* clinical signs or symptoms of heart disease
* hypertension
* coronary disease
* diabetes
* other neurological disease
* cancer
* recent weight change >15 pounds
* abnormal resting ECG
* pregnant and/or breastfeeding women
* underweight and obese individuals (body mass index between 18.5 and 29.9)
* use of amphetamines (Ritalin, Adderall, Concerta) in the past 48 hours
* tibial fracture or tibial stress fracture in the past year
* those with SCI will have no extreme spasticity to avoid spontaneous contractions
* use of baclofen for those with SCI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. A Taylor, PhD, Principal Investigator — Harvard Medical School/Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Cambridge/ Cardiovascular Laboratory, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] BROOKES M. Femoral growth after occlusion of the principal nutrient canal in day-old rabbits. J Bone Joint Surg Br. 1957 Aug;39-B(3):563-71. doi: 10.1302/0301-620X.39B3.563. No abstract available. PMID 13463047
- [Background] Laroche M, Moulinier L, Leger P, Lefebvre D, Mazieres B, Boccalon H. Bone mineral decrease in the leg with unilateral chronic occlusive arterial disease. Clin Exp Rheumatol. 2003 Jan-Feb;21(1):103-6. PMID 12673899
- [Background] Portal-Nunez S, Lozano D, Esbrit P. Role of angiogenesis on bone formation. Histol Histopathol. 2012 May;27(5):559-66. doi: 10.14670/HH-27.559. PMID 22419020
- [Background] Kanczler JM, Oreffo RO. Osteogenesis and angiogenesis: the potential for engineering bone. Eur Cell Mater. 2008 May 2;15:100-14. doi: 10.22203/ecm.v015a08. PMID 18454418
- [Background] Caulkins C, Ebramzadeh E, Winet H. Skeletal muscle contractions uncoupled from gravitational loading directly increase cortical bone blood flow rates in vivo. J Orthop Res. 2009 May;27(5):651-6. doi: 10.1002/jor.20780. PMID 19016540
- [Background] Stabley JN, Moningka NC, Behnke BJ, Delp MD. Exercise training augments regional bone and marrow blood flow during exercise. Med Sci Sports Exerc. 2014 Nov;46(11):2107-12. doi: 10.1249/MSS.0000000000000342. PMID 24658222
- [Background] Stabley JN, Prisby RD, Behnke BJ, Delp MD. Chronic skeletal unloading of the rat femur: mechanisms and functional consequences of vascular remodeling. Bone. 2013 Dec;57(2):355-60. doi: 10.1016/j.bone.2013.09.003. Epub 2013 Sep 19. PMID 24056176
- [Background] Gross PM, Heistad DD, Marcus ML. Neurohumoral regulation of blood flow to bones and marrow. Am J Physiol. 1979 Oct;237(4):H440-8. doi: 10.1152/ajpheart.1979.237.4.H440. PMID 495729
- [Background] Ye Z, Wood MB, Vanhoutte PM. Alpha-adrenergic receptor responsiveness in vascular smooth muscle of canine bone. Clin Orthop Relat Res. 1993 Feb;(287):286-91. PMID 8095442
- [Background] Briggs PJ, Moran CG, Wood MB. Actions of endothelin-1, 2, and 3 in the microvasculature of bone. J Orthop Res. 1998 May;16(3):340-7. doi: 10.1002/jor.1100160310. PMID 9671929
- [Background] Draghici AE, Potart D, Hollmann JL, Pera V, Fang Q, DiMarzio CA, Andrew Taylor J, Niedre MJ, Shefelbine SJ. Near infrared spectroscopy for measuring changes in bone hemoglobin content after exercise in individuals with spinal cord injury. J Orthop Res. 2018 Jan;36(1):183-191. doi: 10.1002/jor.23622. Epub 2017 Jun 28. PMID 28561268
- [Derived] Draghici AE, Ely MR, Hamner JW, Taylor JA. Nitric oxide-mediated vasodilation in human bone. Microcirculation. 2024 Feb;31(2):e12842. doi: 10.1111/micc.12842. Epub 2023 Dec 22. PMID 38133925

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The current study does not assign participants to arms; it is a cross-sectional assessment where all participants will undergo the same procedures. Upon enrollment, all participants underwent laboratory based assessments.
Period: Overall Study
Arm/Group | Laboratory Based Assessments
Started | 90 (Note that the current study as initially approved by the local MGB IRB was not a clinical trial. Once the study was funded, the funding agency NIH/NIAMS requested that the study be designed and registered as a clinical trial. Thus, the initial start date (5/31/2018) was considered the start date of the first enrollment under the approved IRB and not just for the participants enrolled under the NIAMS funding. The date was changed in the protocol section to reflect first enrollment (5/31/2018).)
Completed | 81
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Groups:
- Laboratory Based Assessments: The current study has no arms; it is a cross-sectional assessment where all participants will undergo the same procedures.
  Laboratory based assessments: this is a cross-sectional study including physical maneuvers to assess physiological responses in bone blood flow in young healthy adults and adults with spinal cord injury.
Arm/Group | Laboratory Based Assessments
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants] — Population: Overall number (81) includes both uninjured controls (67) and spinal cord injured individuals (14)
  Participants
    Uninjured controls: number analyzed (Participants) | 67
    Uninjured controls: <=18 years | 0
    Uninjured controls: Between 18 and 65 years | 67
    Uninjured controls: >=65 years | 0
    Spinal cord injury individuals: number analyzed (Participants) | 14
    Spinal cord injury individuals: <=18 years | 0
    Spinal cord injury individuals: Between 18 and 65 years | 14
    Spinal cord injury individuals: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The overall number (81) includes both uninjured controls (67) and spinal cord injured individuals (14).
  Participants
    Uninjured controls: number analyzed (Participants) | 67
    Uninjured controls: Female | 30
    Uninjured controls: Male | 37
    Spinal cord injury individuals: number analyzed (Participants) | 14
    Spinal cord injury individuals: Female | 1
    Spinal cord injury individuals: Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall number (81) includes uninjured controls (67) and spinal cord injured individuals (14).
  Participants
    Uninjured controls: number analyzed (Participants) | 67
    Uninjured controls: Hispanic or Latino | 5
    Uninjured controls: Not Hispanic or Latino | 60
    Uninjured controls: Unknown or Not Reported | 2
    Spinal cord injured individuals: number analyzed (Participants) | 14
    Spinal cord injured individuals: Hispanic or Latino | 2
    Spinal cord injured individuals: Not Hispanic or Latino | 11
    Spinal cord injured individuals: Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall number (81) includes uninjured controls (67) and spinal cord injured individuals (14).
  Participants
    Uninjured controls: number analyzed (Participants) | 67
    Uninjured controls: American Indian or Alaska Native | 1
    Uninjured controls: Asian | 7
    Uninjured controls: Native Hawaiian or Other Pacific Islander | 0
    Uninjured controls: Black or African American | 1
    Uninjured controls: White | 50
    Uninjured controls: More than one race | 1
    Uninjured controls: Unknown or Not Reported | 7
    Spinal cord injured individuals: number analyzed (Participants) | 14
    Spinal cord injured individuals: American Indian or Alaska Native | 0
    Spinal cord injured individuals: Asian | 1
    Spinal cord injured individuals: Native Hawaiian or Other Pacific Islander | 0
    Spinal cord injured individuals: Black or African American | 1
    Spinal cord injured individuals: White | 11
    Spinal cord injured individuals: More than one race | 1
    Spinal cord injured individuals: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Uninjured controls | 67
  United States: Spinal cord injury individuals | 14
Population [Count of Participants; unit: Participants]
  Uninjured controls | 67
  Spinal cord injury individuals | 14
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: The overall number (81) includes uninjured controls (67) and spinal cord injured individuals (14).
  kg/m^2
    Uninjured controls: number analyzed (Participants) | 67
    Uninjured controls | 23.1 (2.9)
    Spinal cord injury individuals: number analyzed (Participants) | 14
    Spinal cord injury individuals | 23.6 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Tibial Blood Perfusion
Description: Concentration of hemoglobin content assessed in response to several physical maneuvers (isometric handgrip exercise, cold pressor test, nitroglycerin, reactive hyperemia, leg dependency). Results are reported in tibial total hemoglobin content (μM). To date there are no absolute established values of tibial bone hemoglobin content and thus an absolute range (minimum and maximum) cannot be provided.
Time Frame: 1 day
Population: 81 participants include 67 controls and 14 SCI across 2 protocols. Thus, most individuals completed only a subset of the total physiological maneuvers.
  After quality control, unusable data was discarded and outcome measures are reported only in the subgroup of individuals (# of participants analyzed for each group included for each test below) analyzed with appropriate data. Reasons for unusable data: spasticity (SCI), unable to complete certain physiological stimuli, motion artifacts.
Measure: Mean (Standard Deviation); unit: μM (concentration)
Arm/Group | Laboratory Based Assessments
Number analyzed (Participants) | 81
μM (concentration)
  Spinal Cord Injury: Isometric handgrip exercise - maximum tibial total hemoglobin (N=14 analyzed): number analyzed (Participants) | 14
  Spinal Cord Injury: Isometric handgrip exercise - maximum tibial total hemoglobin (N=14 analyzed) | 0.54 (1.66)
  Uninjured controls: Isometric handgrip exercise - maximum tibial total hemoglobin (N=13 analyzed): number analyzed (Participants) | 13
  Uninjured controls: Isometric handgrip exercise - maximum tibial total hemoglobin (N=13 analyzed) | -1.47 (3.86)
  Uninjured controls: Cold pressor test - maximum tibial total hemoglobin (N=13 analyzed): number analyzed (Participants) | 13
  Uninjured controls: Cold pressor test - maximum tibial total hemoglobin (N=13 analyzed) | 0.43 (2.18)
  Uninjured controls: Nitroglycerin response - maximum tibial total hemoglobin(N=16 analyzed): number analyzed (Participants) | 16
  Uninjured controls: Nitroglycerin response - maximum tibial total hemoglobin(N=16 analyzed) | 2.08 (0.88)
  Uninjured controls: Reactive hyperemia - maximum tibial total hemoglobin (N=11 analyzed): number analyzed (Participants) | 11
  Uninjured controls: Reactive hyperemia - maximum tibial total hemoglobin (N=11 analyzed) | 3.42 (2.06)
  Uninjured controls: Leg dependency - tibial total hemoglobin (N=14 analyzed): number analyzed (Participants) | 14
  Uninjured controls: Leg dependency - tibial total hemoglobin (N=14 analyzed) | 1.55 (8.55)

ADVERSE EVENTS:
Time Frame: Adverse Events Time Frame - 1 week following study completion.
Arm/Group | Laboratory Based Assessments
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 0/81

LIMITATIONS AND CAVEATS:
This represented an exploratory study of physiological mechanisms underlying bone blood flow regulation in humans. Given the exploratory nature of this work, several technical challenges resulted in unreliable or uninterpretable data which was not included in the final results reported. Technical difficulties included motion artifacts for total hemoglobin measurements, spasticity in adults with spinal cord injury, and inability to perform certain physiological stimuli.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT04083794/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT04083794/ICF_001.pdf